CLINICAL TRIAL: NCT03202056
Title: Effects of Dry Needling Technique in Hip Muscles in Subjects With Grade I-III Hip Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Luis Ceballos Laita, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.I.PI17/0182
Record Dates: First submitted 2017-06-13; First posted 2017-06-28 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Hip Osteoarthritis
Keywords: hip osteoarthritis; physiotherapy; manual therapy
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry needling (Experimental): Dry needling technique in each active myofascial trigger point once per week for 3 weeks.
  Interventions: Other: Dry needling
- Sham Dry needling (Sham Comparator): Sham Dry needling technique in each active myofascial trigger point once per week for 3 weeks.
  Interventions: Other: Sham Dry needling
- Control (No Intervention): Control group. No intervention.

INTERVENTIONS:
Other: Dry needling — Dry needling is a skilled intervention that uses a thin filiform needle to penetrate the skin and stimulate underlying myofascial trigger points, muscular, and connective tissues for the management of neuromusculoskeletal pain and movement impairments.
  Arms: Dry needling
Other: Sham Dry needling — Sham Dry needling use a non-penetrating acupuncture needle
  Arms: Sham Dry needling

SUMMARY:
Dry needling is a new treatment technique, addressed to mechanical pain of the neuromusculoskeletal system. Recent investigations has developed new hypothesis about the etiology of the osteoarthritis and could be in relation to musculoskeletal disorders, but there is no published studies evaluating the results of this technique in hip osteoarthritis patients.

The objective of this trial is to evaluate if dry needling is more effective in symptoms, function, range of motion, strength, muscular length, pain threshold and compared to sham dry needling and control.

For this purpose the investigators conduct a randomized controlled trial double-blind (patient and examiner). The investigators included patients diagnosed of hip osteoarthritis Grade I-III by Scale of Kellgren and Lawrence.

Patients included are randomized into 3 groups one receive Dry needling, other sham dry needling and the other is a control. Groups receive 3 treatment sessions.

The variables are measured at the beginning and end of treatment. And also some variables are measured before and after each session. Patients who participated in sham dry needling or control group, when the intervention finish the investigators will be given the opportunity to receive the actual technique.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed medically with a X-Ray test
* American College of Rheumatology Criteria

Exclusion Criteria:

* Secondary osteoarthritis by a traumatism, Paget disease, inflammatory or metabolic disease, congenital diseases etc.
* Vascular or neurological disease.
* Musculoskeletal pathologies in lumbar spine, pelvis or lower limbs
* Grade IV in Kellgren and Laurence Scale
* Fear of needles

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity with functional tests | Baseline
  The investigators measure the functional capacity with functional test: "test Up and Go" (TUG), "20 and 40 meters self-placed" and "30 seconds-chair stand" at baseline
Intensity symptoms | Baseline
  The investigators measure the intensity of with a visual analogic scale pre-intervention at baseline
Intensity symptoms | through study completion, an average 21 days
  The investigators measure the intensity of with a visual analogic scale at the end of the intervention (3 weeks after baseline the investigators measure the intensity of symptoms through study completion, an average 21 days)
Functional Capacity with functional tests | through study completion, an average 21 days
  The investigator measure the functional capacity with functional test: "Test Up and Go" (TUG test), "20 and 40 meters self-placed" and "30 seconds-chair and stand" at the end of the intervention (through study completion, an average 21 days).

SECONDARY OUTCOMES:
Hip Range of motion | Baseline
  The investigators measure the hip range of motion with an inclinometer at baseline
Hip Range of motion | through study completion, an average 21 days
  The investigators measure the hip range of motion with an inclinometer at the end of the intervention (through study completion, an average 21 days)
Muscular strength | Baseline
  The investigators measure the hip strength with a hand held dynamometer (Lafayette) at baseline
Muscular strength | through study completion, an average 21 days
  The investigators measure the hip strength with a hand held dynamometer (Lafayette) at the end of the intervention (through study completion, an average 21 days)
Muscular length | Baseline
  The investigators measure the muscular length with Passive Knee Extension test, ELY test, and modified Ober test at baseline
Muscular length | through study completion, an average 21 days
  The investigators measure the muscular length with Passive Knee Extension test, ELY test, and modified Ober test at the end of the intervention (through study completion, an average 21 days)
Pain threshold | Baseline
  The investigators measure the pain threshold with a digital algometer in myofascial trigger points of the hip muscles, and also other bone areas to discriminate a central sensitization at baseline
Pain threshold | through study completion, an average 21 days
  The investigators measure the pain threshold with a digital algometer in myofascial trigger points of the hip muscles, and also other bone areas to discriminate a central sensitization at the end of the intervention (through study completion, an average 21 days)
Anxiety and depression with a validated questionnaire (HADS) | Baseline
  The investigators measure the anxiety and depression with HADS questionnaire at baseline
Anxiety and depression with a validated questionnaire (HADS) | through study completion, an average 21 days
  The investigators measure the anxiety and depression with HADS questionnaire at the end of the intervention (through study completion, an average 21 days)
Functional capacity with a validated questionnaire (WOMAC) | Baseline
  The investigator measure the functional capacity with WOMAC questionnaire at baseline
Functional capacity with a validated questionnaire (WOMAC) | through study completion, an average 21 days
  The investigator measure the functional capacity with WOMAC questionnaire at the end of the intervention (through study completion, an average 21 days)
Gait in treadmill | Baseline
  The investigator measure gait pattern in treadmill using wearable inertial sensors to track body kinematics during gait
Gait in treadmill | through study completion
  The investigator measure gait pattern in treadmill using wearable inertial sensors to track body kinematics during gait

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Ceballos Laita, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
The patient data were confidential and were assigned a number to each patient to maintain confidentiality

REFERENCES:
- [Derived] Ceballos-Laita L, Jimenez-Del-Barrio S, Marin-Zurdo J, Moreno-Calvo A, Marin-Bone J, Albarova-Corral MI, Estebanez-de-Miguel E. Effects of dry needling in HIP muscles in patients with HIP osteoarthritis: A randomized controlled trial. Musculoskelet Sci Pract. 2019 Oct;43:76-82. doi: 10.1016/j.msksp.2019.07.006. Epub 2019 Jul 24. PMID 31352178